CLINICAL TRIAL: NCT01282294
Title: Prospective Open Label Post Market Clinical Follow-up to Evaluate the Clinical Usefulness of the Operative Stabilization of Closed and Open Fractures of the Tibia Using Gentamicin - Coated Titanium Nails
Brief Title: Clinical Follow-up to Evaluate the Clinical Usefulness of Gentamicin-coated Titanium Nails in Tibia Fractures
Status: Completed | Type: Observational
Sponsor: Synthes GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: STU-BIO-T-XX-190-02
Record Dates: First submitted 2011-01-21; First posted 2011-01-24 (Estimated); Results first posted 2015-02-11 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-02

CONDITIONS: Tibia Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ETN PROtect: There is only 1 cohort in this case series
  Interventions: Device: ETN PROtect

INTERVENTIONS:
Device: ETN PROtect — Expert Tibial Nail PROtect with Gentamicin coating

SUMMARY:
This post market clinical follow-up is to confirm the clinical usefulness of the Expert Tibial Nail (ETN) PROtect device for operative stabilization in patients with a tibia fracture as measured by the quality of life (EQ5D, SF-12) instruments, disease-specific questionnaires (Iowa Ankle Score, WOMAC) and assessment of (Non-)Device Related Adverse Events or complications.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or more
* Open or closed tibia fracture according to the surgical technique

Exclusion Criteria:

* Women who are pregnant or breast-feeding or are planning to become pregnant during the study
* Patients with consumptive/ malignant primary disease and a life expectancy of < 3 months
* Patients with a known allergy to aminoglycosides
* Physical or mental incapacity, which makes it impossible to obtain informed consent
* History of drug and alcohol abuse
* Patient unlikely to cooperate
* Legal incompetence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the ER with a tibia fracture
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-02; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Raschke, MD, Principal Investigator — University Hospital of Münster, Germany
Locations (4):
- Germany (4):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Heidelberg, Heidelberg
  - University Hospital of Münster, Münster

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ETN PROtect
Started | 100
Intra-operative | 99
Post-operative | 99
6 Weeks | 95
3 Months | 95
6 Months | 94
12 Months | 86
Completed | 81
Not Completed | 19
Not completed — Lost to Follow-up | 14
Not completed — Screening failure | 1
Not completed — Adverse Event | 1
Not completed — Patient non-compliance | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population consistes of patients with an open or closed tibia fracture who were treated with the ETN PROtect.
Arm/Group | ETN PROtect
Number analyzed (Participants) | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 73
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 97
  Negroid | 1
  Asian | 1
  Other | 0
Region of Enrollment [Number; unit: participants]
  Germany | 99
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.2 (5.2)
Height [Mean (Standard Deviation); unit: cm] | 177.6 (8.6)
Weight [Mean (Standard Deviation); unit: kg] | 82.8 (18.7)
Allergies [Number; unit: participants]
  No or unknown | 74
  Metal | 2
  Gentamicin | 0
  Other | 23
Smoking [Number; unit: participants]
  Yes | 31
  No, quit <= 6 Months ago | 4
  No, quit > 6 Months ago | 19
  No, never smoked | 45
Drinking [Number; unit: participants]
  Never drank | 22
  Drinks small amounts (<3 units/day) | 76
  Drinker | 0
  Ex-drinker | 1
Drugs [Number; unit: participants]
  Never used drugs | 84
  Drug abuser | 0
  Ex-drug abuser | 15
Fracture type [Number; unit: participants] — Patients were divided into two groups of fracture types: (1) traumatic/pathologic fractures and (2) other: patients receiving the ETN PROtect due to revision purposes.
  participants
    traumatic/pathologic | 68
    revision purposes | 31
Fracture type (open or closed) [Number; unit: participants]
  Open | 45
  Closed | 50
  None | 1
  Unknown | 3
Time from injury to surgery for traumatic/pathologic patients [Mean (Standard Deviation); unit: days] — The time-to-surgery was recorded for 67 traumatic/pathologic patients.
  days | 8.7 (28.5)
Time from injury to surgery for revision patients [Mean (Standard Deviation); unit: months] — The time-to-surgery was recorded for 21 revision-patients.
  months | 17.1 (16.5)
Use of systemic antibiotics prophylaxis [Number; unit: participants] — More than one option possible.
  participants
    Pre-Operative | 28
    Peri-Operative | 76
    Post-Operative | 32
    None | 0

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life: SF-12 Physical Component Summary (PCS)
Description: The Short Form (SF)-12 health survey comprises 12 questions related to health and wellbeing over the prior four weeks. The responses to these 12 questions are entered into a standardized algorithm to provide summaries of physical and mental health (i.e., physical composite score [PCS] and mental composite score [MCS]). The summary scores are standardized and normalized such that a score of 50 for either the PCS or MCS corresponds to that of an average, healthy person. A score lower than 50 indicates poorer physical and mental health compared to an average, healthy person.
  It was administered at 3, 6, 12 and 18 months post-operatively.
Time Frame: 3, 6, 12 and 18 months post-operatively
Population: Efficacy is based on the number of patients that were treated with the ETN PROtect according to the protocol. Patients were excluded due to a failure to meet the in-/exclusion criteria (2) and a surgical procedure that was not according to the surgical technique (8).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | ETN PROtect
Number analyzed (Participants) | 89
scores on a scale
  Score at 3 months, n=74 | 36.9 (10.0)
  Score at 6 months, n=82 | 41.2 (9.3)
  Score at 12 months, n=74 | 45.6 (9.1)
  Score at 18 months, n=68 | 44.6 (10.7)

2. Primary Outcome: Quality of Life: SF-12 Mental Component Summary (MCS)
Description: The SF-12 short form health survey comprises 12 questions related to health and wellbeing over the prior four weeks. The responses to these 12 questions are entered into a standardized algorithm to provide summaries of physical and mental health (i.e., physical composite score [PCS] and mental composite score [MCS]). The summary scores are standardized and normalized such that a score of 50 for either the PCS or MCS corresponds to that of an average, healthy person. A score lower than 50 indicates poorer physical and mental health compared to an average, healthy person.
  It was administered at 3, 6, 12 and 18 months post-operatively.
Time Frame: 3, 6, 12 and 18 months post-operatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | ETN PROtect
Number analyzed (Participants) | 89
scores on a scale
  Score at 3 months, n=74 | 52.7 (10.8)
  Score at 6 months, n=82 | 53.2 (10.3)
  Score at 12 months, n=74 | 53.3 (9.9)
  Score at 18 months, n=68 | 53.1 (10.2)

3. Primary Outcome: Quality of Life: EQ-5D
Description: The Euroqol Health Survey (EQ-5D, 3-level) was completed on five dimensions (mobility, self care, usual activities, pain/discomfort and anxiety/depression) to measure health-related quality of life on a scale from 0-1. A higher score indicates better quality of life.
Time Frame: 3, 6, 12 and 18 months post-operatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | ETN PROtect
Number analyzed (Participants) | 89
scores on a scale
  Score at 3 months, n=78 | 0.7 (0.2)
  Score at 6 months, n=83 | 0.8 (0.2)
  Score at 12 months, n=78 | 0.8 (0.2)
  Score at 18 months, n=72 | 0.9 (0.1)

4. Secondary Outcome: Evidence of Anatomic Bone Union According to Johnson Classification
Description: Anatomic bone union was assessed according to Johnson et al.*:
  A0: pseudoarthrosis; A1: unilateral pseudoarthrosis; A2: insufficient unilateral bone mass; A3: contiguous union without hypertrophy; A4: solid union of the fracture site.
  *Johnson EE, Urist MR, Finerman GA. Repair of segmental defects of the tibia with cancellous bone grafts augmented with human bone morphogenetic protein. A preliminary report. Clin.Orthop.Relat Res. 1988;249-57
Time Frame: 12 months
Population: Efficacy is based on the number of patients that were treated with the ETN PROtect according to the protocol. Patients were excluded due to a failure to meet the in-/exclusion criteria (2) and a surgical procedure that was not according to the surgical technique (8).
  For the anatomic bone union at 12 months, data of 78 patients is available.
Measure: Number; unit: participants
Arm/Group | ETN PROtect
Number analyzed (Participants) | 78
participants
  A0 | 4
  A1 | 2
  A2 | 9
  A3 | 11
  A4 | 52

5. Secondary Outcome: Evidence of Economic Bone Union According to Johnson Classification
Description: Economic bone union was assessed according to Johnson et al.*:
  E0: complete invalid; E1: no gainful employment; E2: able to work but did not return to previous occupation; E3: returned to previous occupation on a part-time or limited status; E4: returned to previous occupation without restrictions.
  *Johnson EE, Urist MR, Finerman GA. Repair of segmental defects of the tibia with cancellous bone grafts augmented with human bone morphogenetic protein. A preliminary report. Clin.Orthop.Relat Res. 1988;249-57
Time Frame: 12 months
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | ETN PROtect
Number analyzed (Participants) | 78
participants
  E0 | 3
  E1 | 19
  E2 | 8
  E3 | 8
  E4 | 40

6. Secondary Outcome: Evidence of Functional Bone Union According to Johnson Classification
Description: Functional bone union was assessed according to Johnson et al.*:
  F0: motion at the fracture site; F1: level of pain is the same as before operation but able to perform all daily tasks of living; F2: occasional extremity pain and able to perform activities of daily living; F3: no pain and able to perform all activities except sports; F4: complete recovery, no recurrent episodes of pain, and unrestricted activity.
  *Johnson EE, Urist MR, Finerman GA. Repair of segmental defects of the tibia with cancellous bone grafts augmented with human bone morphogenetic protein. A preliminary report. Clin.Orthop.Relat Res. 1988;249-57
Time Frame: 12 months
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | ETN PROtect
Number analyzed (Participants) | 78
participants
  F0 | 4
  F1 | 1
  F2 | 24
  F3 | 17
  F4 | 32

7. Secondary Outcome: Surgeon's Perceived Satisfaction
Description: Surgeons' perceived satisfaction was assessed on a scale from 0 to 100 (0 = very satisfied, 100 = disappointed).
Time Frame: 6 weeks, 3 and 6 months post-operatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | ETN PROtect
Number analyzed (Participants) | 89
scores on a scale
  Score at 6 weeks, n=84 | 18.2 (15.9)
  Score at 3 months, n=82 | 18.9 (16.8)
  Score at 6 months, n=84 | 14.9 (16.7)

8. Primary Outcome: Functional Outcome: IOWA Ankle Score
Description: The Iowa Ankle Score was administered at baseline (retrospective assessment of pre-trauma condition) as well as at 3, 6, 12 and 18 months post-operatively to measures ankle function across four dimensions (function, freedom from pain, gait, range of motion) on a scale of 0-100, where 100 is assigned to full function.
Time Frame: Baseline, 3, 6, 12 and 18 months post-operatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | ETN PROtect
Number analyzed (Participants) | 89
scores on a scale
  Score at Baseline, n=52 | 86.3 (25.7)
  Score at 3 months, n=77 | 62.9 (20.1)
  Score at 6 months, n=84 | 76.4 (19.6)
  Score at 12 months, n=77 | 81.2 (20.3)
  Score at 18 months, n=73 | 85.2 (18.6)

9. Primary Outcome: Functional Outcome: WOMAC
Description: The Western Ontario and McMaster Universities Arthritis Index (WOMAC) questionnaire was administered at 3, 6, 12 and 18 months post-operatively to assess three dimensions: pain, disability and joint stiffness in the knee.
  Each question is scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). The scores are summed up, with a possible score range of 0-96. A higher score on the WOMAC indicate more functional limitations.
Time Frame: 3, 6, 12 and 18 months post-operatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | ETN PROtect
Number analyzed (Participants) | 89
scores on a scale
  Score at 3 months, n=80 | 29.3 (18.5)
  Score at 6 months, n=84 | 24.6 (19.1)
  Score at 12 months, n=76 | 19.2 (19.5)
  Score at 18 months, n=73 | 18.2 (20.0)

10. Primary Outcome: Infection Adverse Events
Description: Infections at the site of ETN PROtect implantation were classified according to Center for Disease Control (CDC) definition into:
  * superficial incisional surgical site infection (SSI), affecting skin and subcutaneous tissue
  * deep incisional SSI, affecting deep soft tissue
  * organ/ space SSI (Osteomyelitis), affecting joint or bursa
Time Frame: 0 - 18 months
Population: as for outcome 1
Measure: Number; unit: number of events
Arm/Group | ETN PROtect
Number analyzed (Participants) | 89
number of events
  superficial incisional SSI at site of ETN PROtect | 6
  deep incisional SSI at site of ETN PROtect | 5
  organ/ space SSI at site of ETN PROtect | 0

11. Secondary Outcome: Likelihood to Develop Wound Infection Assessed by Surgeon
Description: The likelihood to develop a wound infection was assessed by the surgeon on a scale from 0 to 100 (0 = almost nil, 100 = absolutely sure).
Time Frame: 6 weeks, 3 and 6 months post-operatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | ETN PROtect
Number analyzed (Participants) | 89
scores on a scale
  Score at 6 weeks, n=84 | 19.6 (19.6)
  Score at 3 months, n=82 | 14.6 (13.1)
  Score at 6 months, n=84 | 14.4 (19.1)

12. Secondary Outcome: Likelihood to Develop a Non-union Assessed by Surgeon
Description: The likelihood to develop a non-union was assessed by the surgeon on a scale from 0 to 100 (0 = almost nil, 100 = absolutely sure).
Time Frame: 6 weeks, 3 and 6 months post-operatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | ETN PROtect
Number analyzed (Participants) | 89
scores on a scale
  Score at 6 weeks, n=84 | 26.4 (19.1)
  Score at 3 months, n=82 | 23.0 (17.7)
  Score at 6 months, n=84 | 19.6 (21.5)

13. Secondary Outcome: Pain by Visual Analog Scale (VAS)
Description: Leg pain intensity was rated on a 100-mm visual analog scale (VAS). A score of zero indicated no pain at all, and 100 represented the worst possible pain.
Time Frame: 6 weeks, 3, 6, 12 and 18 months post-operatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | ETN PROtect
Number analyzed (Participants) | 89
scores on a scale
  Score at 6 weeks, n=82 | 19.3 (17.4)
  Score at 3 months, n=81 | 24.3 (16.2)
  Score at 6 months, n=84 | 27.0 (21.2)
  Score at 12 months, n=78 | 21.0 (16.3)
  Score at 18 months, n=73 | 23.0 (19.3)

14. Secondary Outcome: Patient's Perceived Satisfaction
Description: Patient's perceived satisfaction was scored on a 100mm visual analog scale (VAS). A score of zero indicated no satisfaction, while a score of 100 indicated completely satisfied.
Time Frame: 6 months
Population: Efficacy is based on the number of patients that were treated with the ETN PROtect according to the protocol. Patients were excluded due to a failure to meet the in-/exclusion criteria (2) and a surgical procedure that was not according to the surgical technique (8).
  Patient satisfaction was completed by 84 patients.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | ETN PROtect
Number analyzed (Participants) | 84
scores on a scale | 63.8 (26.7)

15. Secondary Outcome: Time to Full Weight Bearing
Description: The time from surgery to full weight bearing was assessed in days.
Time Frame: 0 - 18 months
Population: Efficacy is based on the number of patients that were treated with the ETN PROtect according to the protocol. Patients were excluded due to a failure to meet the in-/exclusion criteria (2) and a surgical procedure that was not according to the surgical technique (8). 3 patients never reached full weight bearing, and 1 dropped out before 6 weeks.
Measure: Median (Full Range); unit: days
Arm/Group | ETN PROtect
Number analyzed (Participants) | 85
days | 90.0 [41.0 to 393.0]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from treatment (implantation of the device) through the end of the follow-up period at 18 months.
Arm/Group | ETN PROtect
Serious Adverse Events (participants affected / at risk) | 38/99
Other Adverse Events (participants affected / at risk) | 49/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ETN PROtect (N=99)
BACK PAIN AGGRAVATED (Musculoskeletal and connective tissue disorders) | 1 (1)
COXARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1)
DEVICE BREAKAGE (General disorders) | 2 (2)
DISORDERS OF MUSCLE, LIGAMENT, AND FASCIA (Musculoskeletal and connective tissue disorders) | 1 (1)
ECTOPIC OSSIFICATION (Musculoskeletal and connective tissue disorders) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (1)
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
FISTULA (Musculoskeletal and connective tissue disorders) | 3 (3)
FRACTURE DELAYED UNION (Musculoskeletal and connective tissue disorders) | 5 (6)
FRACTURE MALUNION (Musculoskeletal and connective tissue disorders) | 1 (1)
FRACTURE NONUNION (Musculoskeletal and connective tissue disorders) | 2 (2)
HAMMER TOE (Musculoskeletal and connective tissue disorders) | 1 (1)
HEART ATTACK (Cardiac disorders) | 1 (2)
HEMATOMA (Vascular disorders) | 1 (1)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1)
LOCAL SWELLING (General disorders) | 1 (1)
LOCALIZED INFECTION (Infections and infestations) | 3 (3)
LOSS OF RANGE OF MOTION ASSOCIATED WITH DEVICE (General disorders) | 1 (1)
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
MEDICAL DEVICE COMPLICATION (General disorders) | 1 (1)
NONUNION OF FRACTURE (Musculoskeletal and connective tissue disorders) | 5 (5)
OSTEOMYELITIS (Infections and infestations) | 1 (1)
PAIN IN FOOT (Musculoskeletal and connective tissue disorders) | 1 (1)
PERIPROSTHETIC FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1)
POST-OPERATIVE WOUND INFECTION (Infections and infestations) | 1 (1)
PSEUDARTHROSIS (Musculoskeletal and connective tissue disorders) | 1 (2)
PSYCHOSIS (Psychiatric disorders) | 1 (1)
SKIN NECROSIS (Skin and subcutaneous tissue disorders) | 1 (1)
SOFT TISSUE NECROSIS (Musculoskeletal and connective tissue disorders) | 1 (1)
SURGICAL WOUND INFECTION (Infections and infestations) | 2 (2)
SWELLING (General disorders) | 1 (1)
THROMBOSIS LEG (Vascular disorders) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1)
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 3 (3)
WOUND HEALING DISTURBANCE (General disorders) | 1 (1)
WOUND INFECTION (Infections and infestations) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ETN PROtect (N=99)
ALLERGIC REACTION (Immune system disorders) | 2 (2)
BONE FRACTURE SPONTANEOUS (Musculoskeletal and connective tissue disorders) | 1 (1)
BONE FRAGILE (Musculoskeletal and connective tissue disorders) | 1 (1)
BONE FRAGMENTATION (Injury, poisoning and procedural complications) | 1 (1)
BRONCHITIS (Infections and infestations) | 1 (1)
BRUISE (Injury, poisoning and procedural complications) | 1 (1)
CALF PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
CHONDROPATHY (Musculoskeletal and connective tissue disorders) | 1 (1)
COXARTHROSIS (Musculoskeletal and connective tissue disorders) | 1 (1)
COXITIS (Musculoskeletal and connective tissue disorders) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1)
DEPRESSION WORSENED( (Psychiatric disorders) | 1 (1)
DEPRESSIVE EPISODE (Psychiatric disorders) | 1 (1)
DEVICE POSITIONED INAPPROPRIATELY (General disorders) | 1 (1)
DUODENITIS (Gastrointestinal disorders) | 1 (1)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 (1)
FRACTURE DELAYED UNION (Musculoskeletal and connective tissue disorders) | 2 (2)
GASTRITIS (Gastrointestinal disorders) | 1 (1)
GASTROINTESTINAL INFECTION (Infections and infestations) | 1 (1)
HALLUX VALGUS (Musculoskeletal and connective tissue disorders) | 1 (1)
HEALING DELAYED (General disorders) | 1 (1)
HEMATOMA (Vascular disorders) | 2 (2)
IMPINGEMENT SYNDROME (Musculoskeletal and connective tissue disorders) | 1 (1)
INFLUENZA (Infections and infestations) | 3 (3)
KNEE PAIN (Musculoskeletal and connective tissue disorders) | 4 (4)
LOCAL SWELLING (General disorders) | 1 (1)
LYMPHEDEMA (Vascular disorders) | 2 (2)
NEUROPATHY (Nervous system disorders) | 1 (1)
NON-INSULIN-DEPENDENT DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1)
NONUNION OF FRACTURE (Musculoskeletal and connective tissue disorders) | 1 (1)
NUMBNESS (Nervous system disorders) | 1 (1)
NUMBNESS IN LEG (Nervous system disorders) | 1 (1)
OPERATION SITE BLEED (Injury, poisoning and procedural complications) | 1 (1)
OSTEOMYELITIS (Infections and infestations) | 1 (1)
PAIN (General disorders) | 1 (1)
PAIN IN FOOT (Musculoskeletal and connective tissue disorders) | 1 (1)
PARASTHESIA (Nervous system disorders) | 1 (1)
PATELLAR TENDINITIS (Musculoskeletal and connective tissue disorders) | 1 (1)
PERIPROSTHETIC FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1)
POLYNEUROPATHY (Nervous system disorders) | 1 (1)
PROLONGED POSTTRAUMATIC STRESS DISORDER (Psychiatric disorders) | 1 (1)
SKIN INFECTION (Infections and infestations) | 1 (1)
SKIN LESION NOS (Skin and subcutaneous tissue disorders) | 1 (1)
SKIN NECROSIS( (Skin and subcutaneous tissue disorders) | 1 (1)
STAPHYLOCOCCAL SKIN INFECTION (Infections and infestations) | 1 (1)
STRESS FRACTURE (Injury, poisoning and procedural complications) | 1 (2)
SUBLUXATION PATELLA (Injury, poisoning and procedural complications) | 1 (1)
SURGICAL WOUND INFECTION (Infections and infestations) | 2 (2)
SUTURE GRANULOMA (Injury, poisoning and procedural complications) | 2 (2)
SWELLING (General disorders) | 1 (1)
SWELLING OF LEGS (General disorders) | 1 (1)
TIBIA PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
TOOTHACHE (Gastrointestinal disorders) | 1 (1)
UNEQUAL LEG LENGTH (ACQUIRED) (Musculoskeletal and connective tissue disorders) | 3 (3)
URINARY TRACT DISORDER (Renal and urinary disorders) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1)
WHITLOW (Infections and infestations) | 1 (1)
WOUND HEALING DISTURBANCE (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A single comprehensive publication may be authored on the procedure and outcomes of the trial. Sites that enroll less than five patients will not be included in the publication. Synthes GmbH will have the right to review prior to submission.

Each clinical site that enrolls ten patients will have the option to submit an abstract for publication or presentation at a regional, national, or international conference on their work. Synthes GmbH will have the right to review prior to submission.